CLINICAL TRIAL: NCT03913559
Title: Inotuzumab Ozogamicin for Children With MRD Positive CD22+ Lymphoblastic Leukemia
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Closed due to slow accrual
Sponsor: St. Jude Children's Research Hospital (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INOMRD; NCI-2019-01062 (Registry Identifier: NCI Clinical Trial Registration Program)
Record Dates: First submitted 2019-04-09; First posted 2019-04-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Acute Lymphoblastic Leukemia
Keywords: B-cell Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Burkitt Lymphoma | interventions — Inotuzumab Ozogamicin; Methotrexate; Hydrocortisone; Cytarabine; Diphenhydramine; Acetaminophen; Methylprednisolone; Methylprednisolone Hemisuccinate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Inotuzumab ozogamicin (Experimental): Experimental:Inotuzumab Ozogamicin (InO) Patients with B cell acute lymphoblastic leukemia (B-ALL) that is showing early signs of relapsing (coming back) or is not responding to treatment (refractory).
  Interventions:methotrexate, hydrocortisone and cytarabine into the central nervous system (called triple intrathecal chemotherapy or IT chemotherapy) during this study.
  Premedication: diphenhydramine, acetaminophen and methylprednisolone
  Interventions: Drug: Inotuzumab ozogamicin; Drug: Methotrexate; Drug: Hydrocortisone; Drug: Cytarabine; Drug: Diphenhydramine; Drug: Acetaminophen; Drug: Methylprednisolone

INTERVENTIONS:
Drug: Inotuzumab ozogamicin — dose: 0.5 mg/m2 IV over 60 minutes, days: 1, 8 and 15 every 4 weeks (28 days per cycle) for up to 6 cycles.
  Other Names: Besponsa; CMC-544
Drug: Methotrexate — Intrathecal (IT) therapy
  Other Names: Trexall®
Drug: Hydrocortisone — Intrathecal (IT) therapy
  Other Names: Cortisol
Drug: Cytarabine — Intrathecal (IT) therapy
  Other Names: Ara-C
Drug: Diphenhydramine — 1 mg/kg (max 50 mg) IV
  Other Names: Benadryl
Drug: Acetaminophen — 10 mg/kg (max 650 mg) PO x 1
  Other Names: Tylenol
Drug: Methylprednisolone — 1 mg/kg IV x 1
  Other Names: Solu-Medrol

SUMMARY:
This trial is a limited multi-center, Phase II study to evaluate inotuzumab ozogamicin (Besponsa) in pediatric patients with MRD positive CD22-positive B-lymphoblastic leukemia (B-ALL).

Some patients with newly diagnosed ALL maintain low levels of MRD, despite achieving complete remission with less than 5% blasts in the bone marrow. Others experience re-emergence of low level MRD or increasing levels of MRD on therapy or post-transplant. New approaches are needed to achieve undetectable MRD in these high-risk patients.

Inotuzumab ozogamicin is an antibody-drug conjugate composed of a humanized IgG subtype 4 monoclonal CD22-targeted antibody linked to calicheamicin, a potent anti-tumor antibiotic. CD22 is expressed in more than 90% of patients with B-cell ALL, making it an attractive target in this patient population. Inotuzumab ozogamicin has demonstrated exceptional activity in adults with relapsed or refractory B-ALL.

Primary Objective

* Assess the efficacy of inotuzumab ozogamicin in patients with MRD positive CD22+ B-ALL with 0.1 - 4.99% blasts in bone marrow.

Secondary Objectives

* Study the safety of inotuzumab ozogamicin when used in patients with MRD - positive CD22+ B-ALL with < 5 % blasts in bone marrow.
* Estimate the incidence, severity, and outcome of hepatotoxicity and sinusoidal obstruction syndrome/veno-occlusive disease (SOS/VOD) in patients during inotuzumab ozogamicin and following subsequent treatment, including hematopoietic stem cell transplant (HSCT).

DETAILED DESCRIPTION:
The drug will be administered intravenously on days 1, 8, and 15 of each 28-day cycle. Patients who do not meet the definition of treatment failure after the first cycle may receive up to five additional cycles of therapy. .

After completion of study treatment, patients are followed for 1 year.

ELIGIBILITY:
Inclusion Criteria:

Age

* Participants must be < 22 years of age.

Diagnosis

* Participants must have B-ALL with persistent or rising MRD between 0.1 and 4.99% without extramedullary disease following at least two prior induction attempts, relapse or after hematopoietic stem cell transplant
* Leukemia blasts demonstrating surface expression of CD22

Performance Level

* Karnofsky or Lansky performance score ≥ 50% (corresponding to ECOG Score of ≥ 2). The Lansky performance score should be used for participants < 16 years and the Karnofsky performance score for participants ≥ 16 years.

Prior Therapy

* Patients must have fully recovered from the acute toxic effects of all prior anticancer therapy, defined as resolution of all such toxicities to ≤ Grade 2 or lower per the inclusion/exclusion criteria prior to entering this study.
* At least 14 days must have elapsed since the completion of cytotoxic therapy, with the exception of standard maintenance therapy and steroids.
* At least 7 days must have elapsed since completion of therapy with a biologic agent. For agents that have known adverse events occurring beyond 7 days after administration, this period prior to enrollment must be extended beyond the time during which adverse events are known to occur.
* At least 3 half-lives must have elapsed since prior therapy that included a monoclonal antibody with the exception of blinatumomab. Patients must have been off blinatumomab infusion for at least 7 days and all drug related toxicity must have resolved to Grade 2 or lower as outlined in the inclusion/exclusion criteria.
* At least 42 days must have elapsed since CAR-T cell therapy.
* Participant has received ≤ 1 prior bone marrow transplant.
* At least 90 days have elapsed since bone marrow transplant and participant is off immune suppression for ≥ 2 weeks, if applicable with no evidence of active GVHD.
* At least 2 weeks must have elapsed since local XRT (small port); ≥ 3 months must have elapsed if prior cranial or craniospinal XRT was received, if ≥ 50% of the pelvis was irradiated, or if TBI was received; ≥ 6 weeks must have elapsed if other substantial bone marrow irradiation was given.

Organ Function Requirements

* Adequate renal function defined as glomerular filtration rate ≥ 60 cc/min/1.73m2 or serum creatinine based on age as follows:

  * Age: <6 months; maximum serum creatinine (mg/dL): 0.4 (male, female); Age: 6 months to <1 year; maximum serum creatinine (mg/dL): 0.5 (male, female); Age: 1 to < 2 years; maximum serum creatinine (mg/dL): 0.6 (male, female); Age: 2 to < 6 years; maximum serum creatinine (mg/dL): 0.8 (male, female); Age: 6 to <10 years; maximum serum creatinine (mg/ dL): 1 (male, female); Age: 10 to <13 years; maximum serum creatinine (mg/dL): 1.2 (male, female); Age: 13 to <16 years; maximum serum creatinine (mg/dL): 1.5 (male), 1.4 (female); Age: ≥ 16 years; maximum serum creatinine (mg/dL): 1.7 (male), 1.4 (female)
* Adequate hepatic function defined as:

  * Direct bilirubin ≤ 1.4 mg/dL (if total bilirubin > 1.4 mg/dL) and
  * AST or ALT ≤ 3 x ULN for age.
* Adequate cardiac function defined as shortening fraction of ≥ 27% or ejection fraction ≥ 45%.

Exclusion Criteria:

* History of sinusoidal obstruction syndrome/veno-occlusive disease (SOS/VOD) of any severity.
* Concurrent chemotherapy or targeted anti-cancer agents, other than intrathecal therapy.
* Patient with concurrent severe and/or uncontrolled medical conditions that, in the opinion of the investigator, may impair participation in the study or the evaluation of safety and/or efficacy.
* Known HIV infection or active hepatitis B (defined as hepatitis B surface antigen-positive) or C (defined as hepatitis C antibody-positive).
* Pregnant or lactating (female participant of childbearing potential must have negative serum or urine pregnancy test required within 7 days prior to start of treatment).
* Male or female participant of reproductive potential must agree to use appropriate methods of contraception for the duration of study treatment and for at least 30 days after last dose of protocol treatment.
* Inability or unwillingness of research participant or legal guardian/representative to give written informed consent.

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 5 (Actual)
Dates: Start 2019-05-14 (Actual); Primary Completion 2025-09-15 (Actual); Study Completion 2025-09-15 (Actual)

PRIMARY OUTCOMES:
Treatment response Cycle1 - count | At the end of cycle 1 (each cycle is 28 days)
  Number of patients that reach MRD negative at the end of cycle 1
Treatment Response Cycle 1 - percentage | At the end of cycle 1 (each cycle is 28 days)
  Percentage of patients that reach MRD negative at the end of cycle 1
Treatment Response Cycle 2 - count | At the end of cycle 2 (each cycle is 28 days)
  Number of patients that reach MRD negative at the end of cycle 2
Treatment Response Cycle 2 - percentage | At the end of cycle 2 (each cycle is 28 days)
  Percentage of patients that reach MRD negative at the end of cycle 2

SECONDARY OUTCOMES:
Occurrence of death - count | up to 30 days from last dose of inotuzumab ozogamicin or up to 30 days post-transplant among the patients who proceed to transplant
  Number of patient deaths that occur at any time during observation on study
Occurrence of death - percentage | up to 30 days from last dose of inotuzumab ozogamicin or up to 30 days post-transplant among the patients who proceed to transplant
  Percentage of patient deaths that occur at any time during observation on study
Occurrence of Veno-occlusive disease (VOD) - count | up to 30 days from last dose of inotuzumab ozogamicin or up to 30 days post-transplant among the patients who proceed to transplant
  Number of patients that develop VOD at any time during observation on study
Occurrence of Veno-occlusive disease (VOD) - percentage | up to 30 days from last dose of inotuzumab ozogamicin or up to 30 days post-transplant among the patients who proceed to transplant
  Percentage of patients that develop VOD at any time during observation on study

CONTACTS AND LOCATIONS:
Overall Officials: Sima Jeha, MD, Principal Investigator — St. Jude Children's Research Hospital
Locations (2):
- United States (2):
  - Rady Children's Hospital San Diego, San Diego, California
  - St. Jude Children's Research Hospital, Memphis, Tennessee

IPD SHARING:
Plan to Share IPD: Yes
Individual participant de-identified datasets containing the variables analyzed in the published article will be made available (related to the study primary or secondary objectives contained in the publication). Supporting documents such as the protocol, statistical analyses plan, and informed consent are available through the CTG website for the specific study. Data used to generate the published article will be made available at the time of article publication. Investigators who seek access to individual level de-identified data will contact the computing team in the Department of Biostatistics (ClinTrialDataRequest@stjude.org) who will respond to the data request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be made available at the time of article publication.
Access Criteria: Data will be provided to researchers following a formal request with the following information: full name of requestor, affiliation, data set requested, and timing of when data is needed. As an informational point, the lead statistician and study principal investigator will be informed that primary results datasets have been requested.

REFERENCES:
- [Derived] Shi Z, Zhu Y, Zhang J, Chen B. Monoclonal antibodies: new chance in the management of B-cell acute lymphoblastic leukemia. Hematology. 2022 Dec;27(1):642-652. doi: 10.1080/16078454.2022.2074704. PMID 35622074
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St.Jude — http://www.stjude.org/protocols